CLINICAL TRIAL: NCT05964400
Title: duoABLE for People With Stroke and Their Caregivers (Feasibility)
Brief Title: duoABLE for People With Stroke and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: duoABLE; AOTFIRG23KRINGLE (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Stroke Ischemic; Stroke Hemorrhagic; Stroke Sequelae
Keywords: lifestyle; physical activity; duoABLE; ABLE; rehabilitation; rehab; occupational therapy; physical therapy; stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- duoABLE (Experimental): Stroke participant-caregiver duos (dyads) will meet with an occupational therapist 12 times (2x/week for 6 weeks, approximately 30 minutes/session) to apply activity monitoring, activity scheduling, collaborative problem solving, self-assessment, and social interdependence to self-selected activities that aim to increase both dyad members' physical activity levels
  Interventions: Behavioral: duoABLE

INTERVENTIONS:
Behavioral: duoABLE — Stroke participant-caregiver duos (dyads) will meet with an occupational therapist 12 times (2x/week for 6 weeks, approximately 30 minutes/session) to apply activity monitoring, activity scheduling, collaborative problem solving, self-assessment, and social interdependence to self-selected activities that aim to increase both dyad members' physical activity levels

SUMMARY:
The goal of this intervention study is to test whether a behavioral program that involves people with stroke and their caregivers is acceptable, safe, and can promote physically active lifestyles using enjoyable activities. Participant duos (person with stroke and their caregiver) will be asked to complete assessments at 2 timepoints, wear an activity tracker, participate in 12 sessions with an occupational therapist, and complete an interview.

ELIGIBILITY:
Inclusion Criteria (Stroke Participants):

* Stroke diagnosed more than 6 months ago
* Are 18 years of age or older
* Report ≥6 hours of sedentary behavior on a typical day OR report engagement in ≤90 minutes of moderate-to-vigorous physical activity in the past week
* Reside in a community-based setting
* Are mobile within their home, with or without an assistive device and without physical assistance
* Are able to identify an eligible caregiver who will engage in assessments and intervention.

Inclusion Criteria (Caregiver Participants):

* Are 18 years of age or older
* Report ≥6 hours of sedentary behavior on a typical day OR report engagement in ≤90 minutes of moderate-to-vigorous physical activity in the past week
* Reside in a community-based setting
* Are mobile within their home, with or without an assistive device and without physical assistance

Exclusion Criteria (Stroke Participants):

* Severe aphasia
* Are currently receiving chemotherapy or radiation treatments for cancer
* Have a medical diagnosis of neurodegenerative disorder (i.e., dementia, Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis, glioblastoma)
* Received inpatient treatment for substance use disorder or psychiatric condition within the past 12 months
* Have a history of skin sensitivity related to adhesives
* Are pregnant or expecting to become pregnant in the next 2 months
* Reside in an institutional setting
* Are currently incarcerated

Exclusion Criteria (Caregiver Participants):

* Have a history of skin sensitivity related to adhesives
* Are currently receiving chemotherapy or radiation treatments for cancer
* Have a medical diagnosis of neurodegenerative disorder (i.e., dementia, Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis, glioblastoma)
* Received inpatient treatment for substance use disorder or psychiatric condition within the past 12 months
* Are pregnant or expecting to become pregnant in the next 2 months
* Reside in an institutional setting
* Are currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction | Score at week 8
  Measured using the Client Satisfaction Questionnaire-8 (CSQ-8)

SECONDARY OUTCOMES:
Change in activity restrictions | Baseline to 8 weeks
  Proportion of activities retained assessed at baseline and 8-weeks by the Activity Card Sort 3
Change in sedentary minutes per day | Baseline to 8 weeks
  Minutes of sedentary time per day, measured using the activPAL micro4 (mean minutes per day determined by 7-day wear protocol) at baseline and week 8.
Change in daily step count | Baseline to 8 weeks
  Count of steps per day, measured using the activPAL micro4 (mean daily step count determined by 7-day wear protocol) at baseline and week 8.
Change in Health-related quality of life | Baseline to 8 weeks
  Change in score on the EuroQoL-5 Dimensions-5 Levels (EQ-5D-5L) measured at baseline and week 8
Adverse event count | Count of adverse events at week 8
  Total count of adverse events over the course of the study based on an adverse events questionnaire completed at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Kringle, PhD, OTR/L, Principal Investigator — University of Minnesota
Locations (1):
- School of Kinesiology, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
There are no current plans to share data with other investigators. Upon the completion of the study, a de-identified dataset that includes questionnaire data, raw and processed activPAL data, and transcribed interview data will be created and stored in the DWELL Laboratory at the University of Minnesota. The PI will consider individual requests for data sharing and provide only the necessary de-identified data upon reasonable request, under a University of Minnesota data use agreement.
Supporting Information: Study Protocol, SAP, ICF